CLINICAL TRIAL: NCT01713621
Title: The Extended Observation Over a Period of 28 Days of the Effects of Single Doses of OZ439 on the Recrudescence of Plasmodium Falciparum Malaria - a PhIIa, Open Label Study in Adult Patients
Brief Title: OZ439 PhIIa Study in Plasmodium Falciparum: Extended Observation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_12_006
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Malaria
Keywords: P. falciparum; malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OZ439 100mg (Experimental): Single dose of 100mg of OZ439 administered as an oral suspension
  Interventions: Drug: OZ439
- OZ439 500mg (Experimental): Single dose of 500mg of OZ439 administered as an oral suspension
  Interventions: Drug: OZ439

INTERVENTIONS:
Drug: OZ439 — OZ439 is a novel synthetic trioxolane antimalarial agent

SUMMARY:
This study aims to investigate the concentration dependent effects of OZ439 on the clearance of P. falciparum parasites in patients, specifically the determination of an in-vivo minimum inhibitory concentration (MIC) of OZ439. Characterisation of PK-PD (Pharmacokinetic-Pharmacodynamic) relationships is essential for rational evidence based dosing. The adaptive investigation of a range of doses will provide the best chance of accurate PK-PD characterisation, allowing the observation of Plasmodium falciparum growth dynamics and the subsequent identification of MIC and MPC (minimum parasiticidal concentration). Additionally the tolerability and pharmacokinetics of OZ439 will be confirmed. The PK/PD relationship between OZ439 exposure and subsequent effects on parasitaemia will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the age of 18 and 60 years, inclusive
2. Body weight between 45 kg and 90 kg inclusive
3. Presence of mono-infection of P. falciparum confirmed by:

   1. Fever, as defined by axillary temperature ≥ 37.5°C or oral/rectal/tympanic temperature ≥ 38°C, or history of fever in the previous 24 hours (history of fever must be documented) and,
   2. Microscopically confirmed parasite infection: 1,000 to 75,000 asexual parasite count/µL blood.
4. Written informed consent, in accordance with local practice, provided by patient. If the patient is unable to write, witnessed consent is permitted according to local ethical considerations
5. Ability to swallow oral medication
6. Ability and willingness to participate and access the health facility
7. Agree to hospitalization for at least 72h until parasites have fallen below the level of polymerase chain reaction (PCR) detection and have no signs or symptoms of malaria; and then to return once daily to the study centre for blood sampling for quantitative polymerase chain reaction (qPCR), and rehospitalisation when qPCR levels are detectable.

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment according to the World Health Organization Criteria 2010
2. Mixed Plasmodium infection
3. Severe vomiting, defined as more than three times in the 24 hours prior to inclusion in the study or inability to tolerate oral treatment, or severe diarrhoea defined as 3 or more watery stools per day
4. Presence of other serious or chronic clinical condition requiring hospitalization
5. Severe malnutrition (defined as the weight-for-height being below -3 standard deviation or less than 70% of median of the NCHS/WHO normalized reference values)
6. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, QTc interval greater than or equal to 450 msec), respiratory (including active tuberculosis), history of jaundice, hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric, history of convulsions or other abnormality (including head trauma)
7. Known history of hypersensitivity, allergic or adverse reactions to artemisinin containing compounds or mefloquine
8. Known active Hepatitis A Immunoglobulin M (IgM) (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab)
9. Have received any antimalarial treatment in the preceding 14 days, as determined by history and screening test
10. Have received antibacterial with known antimalarial activity in the preceding 14 days
11. Have received an investigational drug within the past 4 weeks
12. Liver function tests (Aspartate Aminotransferase(ASAT)/Alanine Aminotransferase (ALAT) levels) > 2x upper limit of normal (ULN) if Total Bilirubin normal or >1.5xULN if Total bilirubin between >1 and >1.5xULN
13. Hemoglobin (Hb) level =< 8g/dl
14. Total Bilirubin > 1.5XULN
15. Serum creatinine levels more than 2 times the upper limit of normal range (>2xULN).
16. Female patients must be neither pregnant as demonstrated by a negative serum pregnancy test at screening and urinary pregnancy test pre-dose (the result of the pre-dose assessment must be confirmed negative prior to dosing) nor lactating, and must be willing to take measures not to become pregnant during the study period and safety follow-up period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sasithon Pukrittayakamee, MD, Principal Investigator — Faculty of Tropical Medicine, Mahidol University, Bangkok; Francois Nosten, MD, Principal Investigator — Shoklo Malaria Research Unit, Faculty of Tropical medicine, Mahidol University
Locations (3):
- Thailand (3):
  - Faculty of Tropical Medicine,, Bangkok, Bangkok
  - Mae Ramat District hospital, Mae Ramat, Changwat Tak
  - Shoklo Malaria Research Unit, Mae Sot, Changwat Tak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vennerstrom JL, Arbe-Barnes S, Brun R, Charman SA, Chiu FC, Chollet J, Dong Y, Dorn A, Hunziker D, Matile H, McIntosh K, Padmanilayam M, Santo Tomas J, Scheurer C, Scorneaux B, Tang Y, Urwyler H, Wittlin S, Charman WN. Identification of an antimalarial synthetic trioxolane drug development candidate. Nature. 2004 Aug 19;430(7002):900-4. doi: 10.1038/nature02779. PMID 15318224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited and followed up over 28 days in four clinics in Thailand from April 2013 to April 2015.
Period: Overall Study
Arm/Group | OZ439 100mg | OZ439 500mg
Started | 8 | 17
Completed | 1 | 1
Not Completed | 7 | 16

BASELINE CHARACTERISTICS:
Population: Analysed:
  Safety population: 25 patients Intent to Treat population: 23 patients Per Protocol population: 22 patients
  Pharmacokinetic (PK) population:
  Noncompartmental PK Analysis:19 patients Population PK Analysis: 22 patients
Groups:
- Total: Total of all reporting groups
Arm/Group | OZ439 100mg | OZ439 500mg | Total
Number analyzed (Participants) | 8 | 17 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12.44) | 34 (10.49) | 35 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 7 | 14 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 17 | 25
Region of Enrollment [Number; unit: participants]
  Thailand | 8 | 17 | 25

OUTCOME MEASURES:

1. Primary Outcome: Minimum Inhibitory Concentration (MIC) and Minimum Parasiticidal Concentration (MPC)
Description: The estimated MIC and MPC were derived from the fitted parasitaemia concentration and PK/PD relationship.
Time Frame: up to 28 days
Population: Model predicted MIC and MPC
Measure: Mean (Standard Deviation); unit: ng/Ml
Arm/Group | OZ439 100mg | OZ439 500mg
Number analyzed (Participants) | 7 | 15
ng/Ml
  Model predicted MIC | 2.4 (3.5) | 4.1 (5)
  Model predicted MPC | 77 (128) | 319 (877)

ADVERSE EVENTS:
Time Frame: Patients were assessed for AEs for the duration of the study during the extended observation period, until study discontinuation and the follow-up visit.
Arm/Group | OZ439 100mg | OZ439 500mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/17
Other Adverse Events (participants affected / at risk) | 6/8 | 10/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OZ439 100mg (N=8) | OZ439 500mg (N=17)
vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (3) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (2) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 2 (2) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
LEUKOCYTURIA (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less